CLINICAL TRIAL: NCT00001904
Title: Assessment of a B-Mode Ultrasound Technique for the Measurement of Carotid Artery Intima-Media Thickness
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990085; 99-I-0085
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Atherosclerosis; Myocardial Infarction
Keywords: Atherosclerosis; Cardiovascular Disease; Computerized Edge Reader; Myocardial Infarction; Risk Factor
MeSH Terms: conditions — Atherosclerosis; Myocardial Infarction; Cardiovascular Diseases

SUMMARY:
This minimal risk protocol is designed to assess the reproducibility of B-mode ultrasound measurements of carotid intima media thickness (IMT) when the scans are performed in CC Radiology and read using a computerized edge reader. Up to 20 volunteers will have two ultrasounds performed within a 6-month period. IMT thickness is used as a surrogate marker for atherosclerosis and may be of value in clinical trials.

DETAILED DESCRIPTION:
This minimal risk protocol is designed to assess the reproducibility of B-mode ultrasound measurements of carotid intima-media thickness (IMT) when the scans are performed in CC Radiology and read using a computerized edge reader. Up to 50 volunteers will have two ultrasounds performed within a 6-month period. IMT thickness is used as a surrogate marker for atherosclerosis and may be of value in clinical trials.

ELIGIBILITY:
Adult (age 18 or older).

Desire to participate in the study; willing and able to provide informed consent.

No history of stroke or carotid disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1999-04; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Tan GH, Gharib H. Thyroid incidentalomas: management approaches to nonpalpable nodules discovered incidentally on thyroid imaging. Ann Intern Med. 1997 Feb 1;126(3):226-31. doi: 10.7326/0003-4819-126-3-199702010-00009. PMID 9027275
- [Background] Mercuri M. Noninvasive imaging protocols to detect and monitor carotid atherosclerosis progression. Am J Hypertens. 1994 Jul;7(7 Pt 2):23S-29S. doi: 10.1093/ajh/7.7.23s. PMID 7946175